CLINICAL TRIAL: NCT02707575
Title: Cytokeratin 8 Level in Aqueous Humor, as a Prognostic Factor for Visual and Anatomical Outcomes After Ranibizumab (Lucentis) in Neovascular Age-related Macular Degeneration
Brief Title: Cytokeratin 8 Level in Age-related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Konkuk University (Other); Inje University (Other); Novartis (Industry); Severance Hospital (Other)
Responsible Party: Principal Investigator, Suk Ho Byeon, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2015-0304
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Age-related Macular Degeneration
Keywords: Keratin; Ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ranibizumab: Intravitreal Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Three monthly consecutive injections of 0.5-mg ranibizumab will be performed. Aqueous humor samples will be taken each time an intravitreal injection in indicated and performed.
  Other Names: Lucentis

SUMMARY:
The investigators will evaluate the concentrations of cytokeratin 8 in aqueous humor in eyes with exudative age-related macular degeneration (AMD) before therapy with intravitreal Ranibizumab, and identify associations with visual and anatomical outcome after treatment.

DETAILED DESCRIPTION:
In this non-randomized, and open-label study, the investigators will prospectively evaluate 58 patients with treatment naive exudative age-related macular degeneration (AMD) who receive intravitreal ranibizumab injection. A mean volume of 0.1 ml of aqueous humor samples will be taken each time an intravitreal injection is indicated and performed. Cytokeratin 8 level in aqueous humor will be evaluated, and associations of baseline cytokeratin 8 level and visual (the best corrected visual acuity change) and anatomical (optical coherence tomography parameters) after Ranibizumab injection will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naive neovascular AMD patients requiring intravitreal injection of Ranibizumab
2. A recent onset of disease confirmed by history and clinical findings.
3. Patient is required to be least 50 years of age

Exclusion Criteria:

1. Myopia with a refractive error >-3.0 diopters or evidence of pathologic myopia (pre-operative refractive data were used to assess pseudophakic eyes)
2. Any history of vitrectomy, anti-VEGF therapy, or photodynamic therapy (PDT)
3. History of cataract surgery within 3 months prior to presentation
4. Evidence of end-stage AMD such as subfoveal fibrosis or atrophy
5. Evidence of other retinal diseases including central serous chorioretinopathy and other neovascularmaculopathies; glaucoma; poor imaging data caused by media opacity; or unstable fixation
6. Patients with uncontrolled systemic diseases, use of immunosuppressive drugs, or malignant tumors of any location

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patient is required to be least 50 years of age with newly diagnosed exudative age-related macular degeneration, with a recent onset of disease.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
The changes in the Logarithm of the Minimum Angle of Resolution (LogMAR) visual acuity | From baseline to one month after three monthly consecutive ranibizumab injection
  The changes in the Logarithm of the Minimum Angle of Resolution (LogMAR) visual acuity

SECONDARY OUTCOMES:
The presence of intra/subretinal fluid on Spectral domain (SD)- Optical Coherence Tomography (OCT) | From baseline to one month after three monthly consecutive ranibizumab injection
  The presence of intra/subretinal fluid on Spectral domain (SD)- Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Suk Ho Byeon, MD. Ph.D., Principal Investigator — Professor. Yonsei University
Locations (2):
- South Korea (2):
  - Inje University Ilsan Paik Hospital, Goyang
  - Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT02707575/Prot_SAP_000.pdf